CLINICAL TRIAL: NCT02003261
Title: An Assessor-blinded, Randomized, 20-week, Parallel-group, Superiority Study to Compare the Efficacy of Transdiagnostic Cognitive Behavioral Therapy Versus Waiting-list in Depressive and Anxiety Symptoms of Depressive and Anxiety Disorders
Brief Title: Japan Unified Protocol Clinical Trial for Depressive and Anxiety Disorders (JUNP Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Principal Investigator, Masaya ITO, Chief of dissemination and training at National Center of Cognitive-Behavior Therapy and Research, National Center of Neurology and Psychiatry, Japan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAKENHI 25705018
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Anxiety Disorders; Depressive Disorders
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder | interventions — Therapeutics; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unified Protocol with Treatment As Usual (Experimental): Unified Protocol is designed to help patients learn how to confront and experience uncomfortable emotions and learn how to respond to their emotions in more adaptive ways. Individual treatment sessions will be conducted by experienced clinicians who will be trained in the administration of this protocol. A workbook will be provided to each patient as part of this manualized treatment. During this treatment period, the participants continue the Treatment As Usual.
  Interventions: Behavioral: Unified Protocol with Treatment As Usual; Other: Treatment As Usual
- Waitlist Control with Treatment As Usual (Other): Waitlist participants will not receive treatment during a 20-week waitlist period, but will receive the unified protocol immediately following the 20 week waiting period. During the waitlist period, the waitlist participants continue the treatment as usual.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Unified Protocol with Treatment As Usual — Unified Protocol(UP) is a transdiagnostic cognitive-behavioral therapy for depressive and anxiety disorders, which is developed by Dr. Barlow and his colleagues at Boston university.
  UP is weekly, face to face, individual psychotherapy consisting of 9 to 20 sessions. Average session number is 16 sessions. Contents of the treatment includes motivational enhancement, psychoeducation of treatment rationale and emotion, emotion awareness training, cognitive reappraisal, avoidance and emotion driven behaviors, interoceptive exposure and emotion exposure.
  Other Names: Cognitive Behavioral Therapy
  Arms: Unified Protocol with Treatment As Usual
Other: Treatment As Usual — Most of the TAU will be drug therapy or nonsystematic supportive psychotherapy.

SUMMARY:
This study is to examine the superiority of the combined treatments of transdiagnostic cognitive-behavior therapy (Unified Protocol; UP) and Treatment-As-Usual in comparison with the waiting-list with Treatment-As-Usual in the reduction of depressive and anxiety symptoms among depressive and anxiety disorders.

DETAILED DESCRIPTION:
Participants with depressive or anxiety disorders will be randomized to either Unified Protocol with Treatment-As-Usual or Wail-list with Treatment-As-Usual. Intervention period will be 20-week and the follow-up period will be 43 week from registration.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Major Depressive Disorder, Dysthymia, Depressive Disorder Not Otherwise Specified, Panic Disorder With Agoraphobia, Panic Disorder Without Agoraphobia, Agoraphobia Without History of Panic Disorder, Social Phobia(Social Anxiety Disorder), Obsessive-Compulsive Disorder, Posttraumatic Stress Disorder, Generalized Anxiety Disorder, Anxiety Disorder Not Otherwise Specified assessed by SCID.
* Depressive and anxiety symptoms is mild or more severe (GRID-HAMD >= 8).
* Ages 20 years or older, and 65 years or younger at screening.
* Subjects who give full consent in the participation of the study.

Exclusion Criteria:

* No alcohol or substance use disorder in 6 months prior to the screening assessed by SCID
* No current manic episode or current schizophrenia and other psychotic disorders at baseline assessed by SCID
* No serious suicidal ideation at baseline (GRID-HAMD Item3 severity is 3 or higher.)
* No life-threatening, severe or unstable physical disorders or major cognitive deficits at baseline.
* Evidence of unable to participate half or more of the intervention phase.
* No structured psychotherapy during at baseline.
* Other relevant reason decided by the investigators.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
GRID-Hamilton Depression Rating Scale-17 (GRID-HAMD) | 21 weeks

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale 14 item(HAM-A) | 21 weeks
Clinical Global Impression- Severity(CGI-S) | 21 weeks
Clinical Global Impression-Improvement(CGI-I) | 21 weeks
Responder Status assessed by GRID-HAMD | 21 weeks
  Reduction in GRID-HAMD score of at least 50% compared with baseline
Remission of symptoms assessed by GRID-HAMD | 21 weeks
  GRID-HAMD score of less than 8
Psychiatric diagnosis assessed by Structured Clinical Interview for the DSM(SCID) | 21 weeks

OTHER OUTCOMES:
Global Assessment of Functioning(GAF) | 10 weeks, 21 weeks, and 43 weeks
Disorder specific measures | 10 weeks, 21 weeks, and 43 weeks
  Participants will be answered some of the following measures in accord with their diagnoses; Beck Depression Inventory-II for Depressive Disorders, Panic Disorder Severity Scale for Panic Disorder, Penn-State Worry Questionnaire for Generalized Anxiety Disorder, Impact of Event Scale-Revised for Post-Traumatic Stress Disorder, Yale-Brown Obsessive Compulsive Scale for Obsessive Compulsive Disorder and Fear Questionnaire for Agora Phobia.
Quality of Life(EQ-5D) | 10 weeks, 21 weeks, and 43 weeks
Sheehan Disability Scale(SDISS) | 10 weeks, 21 weeks, and 43 weeks
Sense of Authenticity Scale(SOA) | 10 weeks, 21 weeks, and 43 weeks
Overall Anxiety Severity and Impairment Scale(OASIS) | 10 weeks, 21 weeks, 43 weeks and at every UP sessions
Overall Depression Severity and Impairment Scale(ODSIS) | 10 weeks, 21 weeks, 43 weeks and at every UP sessions
Eysenck Personality Questionnaire- Revised Short version, Neuroticism(EPQR-S) | 10 weeks, 21 weeks, 43 weeks and at UP session #5 and #15
Anxiety Sensitivity Index-III(ASI-III) | 10 weeks, 21 weeks, 43 weeks and at UP session #5 and #15
Emotion Regulation Skills Questionnaire(ERSQ) | 10 weeks, 21 weeks, 43 weeks and at UP session #5 and #15
Credibility/Expectancy Questionnaire(CEQ) | 2 weeks
Session Rating Scale(SRS V.3.0) | UP session at #1, 5, 10, and 15
Homework Compliance Scale(HCS) | UP session at #1, 5, 10, and 15
Adverse Events | From 1 week to 21 weeks
  Adverse Events will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
GRID-Hamilton Depression Rating Scale-17 (GRID-HAMD) | 10 weeks, 43 weeks
Hamilton Anxiety Rating Scale 14 item(HAM-A) | 10 weeks and 43 weeks
Clinical Global Impression- Severity(CGI-S) | 10 weeks, 43 weeks
Clinical Global Impression-Improvement(CGI-I) | 10 weeks, 43 weeks
Psychiatric diagnosis assessed by SCID | 43 weeks
Emotion Exposure Scale (EES) | 10 weeks, 21 weeks, 43 weeks
Understanding of Treatment Rational of Unified Protocol (TRUP) | 10 weeks, 21 weeks, and 43 weeks
Magnetic Resonance Imaging(MRI) | 21 weeks, 43 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Masaya Ito, Ph.D., Principal Investigator — National Center for Cognitive-Behavior Therapy and Research, National Center of Neurology and Psychiatry
Locations (1):
- National Center of Neurology and Psychiatry, Kodaira, Tokyo, Japan

REFERENCES:
- [Derived] Ito M, Okumura Y, Horikoshi M, Kato N, Oe Y, Miyamae M, Hirabayashi N, Kanie A, Nakagawa A, Ono Y. Japan Unified Protocol Clinical Trial for Depressive and Anxiety Disorders (JUNP study): study protocol for a randomized controlled trial. BMC Psychiatry. 2016 Mar 18;16:71. doi: 10.1186/s12888-016-0779-8. PMID 26987315